CLINICAL TRIAL: NCT05581511
Title: Natural History Study of Cutaneous Neurofibromas in People With Neurofibromatosis Type 1
Brief Title: Natural History Study of Cutaneous Neurofibromas in People With NF1
Acronym: cNF Natural Hx
Status: Active, not recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Neurofibromatosis Therapeutic Acceleration Program (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB00272137
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Neurofibromatosis Type 1; Neurofibromatosis 1; Neurofibromatosis (Nonmalignant); Cutaneous Neurofibroma
Keywords: neurofibroma; cutaneous neurofibroma; neurofibromas; cutaneous neurofibromas; skin neurofibromas; dermal neurofibromas; neurofibromatosis; neurofibromatosis type 1; neurofibromatosis 1; von Recklinghausen syndrome; von Recklinghausen disease; NF1
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibromatoses; Neurofibroma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Optional donations of blood and cutaneous neurofibroma are accepted
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluation of the natural history of cutaneous neurofibromas — Cutaneous neurofibromas (cNFs) are the most common tumors in people with neurofibromatosis type 1 (NF1). Despite their benign histology, they can significantly impact patients' quality of life (QoL). In this project, the natural history of cNFs will be prospectively and systematically studied. To accomplish this, the reproducibility and efficiency of using 3D whole-body photography was evaluated in a small cohort of patients. The study is enrolling patients of all ages with cNFs into groups by epochs of life to characterize the baseline tumor burden and the change in number and morphology of cNFs over five years. In addition, the study will perform next generation sequencing to describe the genetic variations in the NF1 gene and evaluate potential relations between genotype and phenotype. Lastly, the study will validate clinician- and patient-reported severity scales of cNFs developed for this patient population.

SUMMARY:
People diagnosed with NF1 may develop cutaneous neurofibromas, also known as cNFs. These benign tumors can cause discomfort and affect a person's quality of life. Researchers at Johns Hopkins are studying how cNF tumors form, grow and change over time. This information may help doctors in the future, provide early interventions and improve quality of life for NF1 patients. Researchers will also explore a new way of monitoring cNF with 3D camera technology. People of all ages with NF1, living in the United States, are invited to participate in this important research study.

DETAILED DESCRIPTION:
The majority of people diagnosed with Neurofibromatosis Type 1 are likely to develop at least one cutaneous neurofibroma-also known as cNF. While benign, these tumors can cause pain, itchiness, disfigurement, and dramatically affect a person's quality of life; and little is known about how it forms and grows. A team of researchers at Johns Hopkins is studying the natural history of cNF to better understand how cNF tumors develop and change over time. This research may help doctors provide early intervention to people at risk of developing cNF, or prevent cNF altogether. And, it will help prioritize future research focused on improving the quality of life for people who have NF1

People of all ages diagnosed with NF1 are invited to participate in this research study. Participants under the age of 18 with parental consent are welcome. Participants will need to provide a saliva sample for genetic testing and NF1 gene identification. Once a year for the next five years, participants will undergo whole-body, 3D imaging. This imaging technology will generate a three-dimensional, digital image with which researchers will monitor changes in cNF over time. It does not use radiation and has no expected side effects.

Participants will need to answer annual health surveys to monitor quality of life, NF1 and cNF symptoms. Participants may also choose to donate blood and tissue samples for future NF research initiatives.

The study is open to anyone with NF1 living in the United States. Annual visits for this study will take place at the Johns Hopkins Outpatient Center in Baltimore, Maryland. There is no cost to the participants, and eligible travel and parking expenses may be reimbursed up to a specified amount. In fact, participants will receive a gift card at the first visit for participating in the study.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of NF1 based on NIH Consensus Conference clinical criteria or confirmed pathogenic NF1 mutation
* Patients ages 1-100 will be eligible to participate
* Ability have 3D whole-body pictures taken which entails standing still for a few seconds
* Ability to provide informed consent or obtain consent from parent or legally authorized representative in the case of patients under 18 years of age who cannot consent for themselves or those with disabilities preventing them from participating in the consent process.
* Participants must be able to travel to Johns Hopkins Hospital for whole-body imaging and physical exam.

Exclusion criteria:

* Concurrent experimental or off label use of therapies for cNF

Ages: 1 Year to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: People of all ages with NF1
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-06-28 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Tumor burden of cutaneous neurofibromas in people with neurofibromatosis type 1 (NF1). | Baseline
  To characterize the baseline tumor burden of cNFs
Change in number of cNFs | Once per year over 5 years
  Change in number of cNFs once per year over five years.

SECONDARY OUTCOMES:
To characterize the genetic variations in the NF1 gene and evaluate potential relations between genotype and phenotype. | 2 years
  Using Next Generation Sequencing (NGS) to evaluate pathogenic variants in the NF1 gene and their relation to cNF tumor burden

CONTACTS AND LOCATIONS:
Overall Officials: Carlos G Romo, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States